CLINICAL TRIAL: NCT06902259
Title: The Effect of Breath Exercıse and Reıkı Applıcatıon on Tıredness and Nausea and Vomiting Management in Oncology Patıents; Randomısed Controlled Study
Brief Title: The Effect of Breath Exercıse and Reıkı Applıcatıon
Acronym: Reiki App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aslıhan ÖZTÜRK ÇETİN (Other)
Responsible Party: Sponsor-Investigator, Aslıhan ÖZTÜRK ÇETİN, Res. Ass. RN, MSc, PhD, Izmir Bakircay University
Organization: Izmir Bakircay University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Bakircay Unversity
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Reiki; Breath Exercise; Tıredness and Nausea and Vomiting Management
Keywords: reiki; symptom management; breath exercise; oncology patients
MeSH Terms: conditions — Nausea

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Sixty patients, including 20 patients in each group, who met the inclusion criteria were identified. The details of the study were explained to the patients and their consent was obtained. In order to minimise selection bias, a simple random sampling method, the random numbers table, was used and patients were assigned to groups as 20 reiki group, 20 breathing exercise group and 20 control group.
- Breathing exercise group (Other): Sixty patients, including 20 patients in each group, who met the inclusion criteria were identified. The details of the study were explained to the patients and their consent was obtained. In order to minimise selection bias, a simple random sampling method, the random numbers table, was used and patients were assigned to groups as 20 reiki group, 20 breathing exercise group and 20 control group.
  Interventions: Other: randomised controlled trial
- Reiki group (Other): Sixty patients, including 20 patients in each group, who met the inclusion criteria were identified. The details of the study were explained to the patients and their consent was obtained. In order to minimise selection bias, a simple random sampling method, the random numbers table, was used and patients were assigned to groups as 20 reiki group, 20 breathing exercise group and 20 control group.
  Interventions: Other: randomised controlled trial

INTERVENTIONS:
Other: randomised controlled trial — Breathing exercise group: Sixty patients, including 20 patients in each group, who met the inclusion criteria were identified. The details of the study were explained to the patients and their consent was obtained. In order to minimise selection bias, a simple random sampling method, the random numbers table, was used and patients were assigned to groups as 20 reiki group, 20 breathing exercise group and 20 control group.
  Reiki group: Sixty patients, including 20 patients in each group, who met the inclusion criteria were identified. The details of the study were explained to the patients and their consent was obtained. In order to minimise selection bias, a simple random sampling method, the random numbers table, was used and patients were assigned to groups as 20 reiki group, 20 breathing exercise group and 20 control group.
  Arms: Breathing exercise group; Reiki group

SUMMARY:
: This randomised controlled trial was conducted to investigate the effects of breathing exercise and reiki on fatigue and nausea and vomiting symptoms in oncology patients. Data were collected between 1 December 2023 and 30 May 2024, just before the patients started chemotherapy treatment, using data collection forms with a face-to-face interview method of approximately 30 minutes. Since it was thought that there might be case losses during the study, it was decided to take 20 patients for both groups.

DETAILED DESCRIPTION:
The study was conducted with cancer patients receiving treatment in the outpatient chemotherapy unit of a university hospital between 1 December 2024 and 30 May 2024.The population of the study was 600 cancer patients receiving chemotherapy in the Outpatient Chemotherapy Unit of a university hospital. The sample consisted of patients who applied to the Medical Oncology Outpatient Clinic for treatment between 1 December 2023 and 30 May 2024, who accepted to participate in the study and met the inclusion criteria. Power analysis was performed to determine the sample size. The power of the study was calculated with the G Power 3.1 programme. Accordingly, it was determined that there should be at least 18 patients in each group. Since it was thought that there might be case losses during the study, it was decided to take 20 patients for both groups. Sixty patients, including 20 patients in each group, who met the inclusion criteria were identified. The details of the study were explained to the patients and their consent was obtained. In order to minimise selection bias, a simple random sampling method, the random numbers table, was used and patients were assigned to groups as 20 reiki group, 20 breathing exercise group and 20 control group.Patients who volunteered to participate in the study, were diagnosed with cancer, had symptoms of nausea-vomiting and fatigue, were literate, could communicate, did not have a diagnosis of mental or psychiatric illness, were not hearing or visually impaired, were 18 years of age or older, and were not receiving antiemetic treatment.

Exclusion criteria: Patients with any other disease related to the gastrointestinal system, any other disease or condition that would prevent them from performing the exercises to be performed for the study.

Before starting the study, approval was obtained from the Bakırçay University Non-Interventional Clinical Research Ethics Committee of a state university (25.10.2023/Decision no: 1259). Institutional permission was obtained from the hospital where the study was conducted. In order to use the Hirai Cancer Fatigue Scale in the study, permission to use the scale was obtained from the author via e-mail. Verbal and written informed consent was obtained from all participants. The study was conducted according to the principles of the Helsinki Declaration of Human Rights.The data obtained in the study were analysed using SPSS (Statistical Package for Social Sciences) for Windows 22.0 software. Number, percentage, mean, standard deviation were used as descriptive statistical methods in the evaluation of the data. Differences between the rates of categorical variables in independent groups were analysed by Chi-Square tests. Kurtosis and Skewness values were analysed to determine whether the research variables showed normal distribution.

In the related literature, the results of kurtosis and skewness values of the variables between +1.5 and -1.5, +2.0 and -2.0 are accepted as normal distribution. Since it was determined that the variables were normally distributed, parametric methods were used to analyse the data [15,16]. One way Anova test was used to compare quantitative continuous data between groups. Scheffe test was used as a complementary post-hoc analysis to determine the differences after the Anova test. Repeated measures ANOVA test and complementary Bonferroni test were used for the comparison of intra-group measurements.

ELIGIBILITY:
Inclusion Criteria:

Patients who volunteered to participate in the study, were diagnosed with cancer, had symptoms of nausea-vomiting and fatigue, were literate, could communicate, did not have a diagnosis of mental or psychiatric illness, were not hearing or visually impaired, were 18 years of age or older, and were not receiving antiemetic treatment.

Exclusion Criteria:

Patients with any other disease related to the gastrointestinal system, any other disease or condition that would prevent them from performing the exercises to be performed for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Individual Introductory Information Form | 4 months
  The Individual Descriptive Information Form was prepared by the researchers in line with the literature information and consists of questions such as socio-demographic characteristics such as age, marital status, chronic diseases, disease history, and type, stage, metastasis status, metastasis site, treatment status, nausea and vomiting [5-9].

SECONDARY OUTCOMES:
Hirai Cancer Fatigue Scale | 4 months
  The scale developed by Kazue Hirai et al. in 2015 and adapted into Turkish by Mencel in 2021 consists of 15 items. The scale measures fatigue in cancer patients and is 5-point Likert type. Each item of the scale is evaluated as 1 'not at all', 2 'very little', 3 'a little', 4 'a lot', 5 'very much'. There are 3 sub-dimensions: physical - mental sub-dimension, activity-related sensitivity, cognitive sensitivity. Items 1-6 in the scale include physical-mental sub-dimension, items 7-12 include activity-related sensitivity sub-dimension and items 12-15 include cognitive sensitivity sub-dimension. The scale has no cut-off point. The minimum value of the scale is 15 and the maximum value is 75. High scores on the scale indicate increased fatigue and low scores indicate decreased fatigue.14 The Cronbach Alpha value of the original scale was found to be 0.943. The Cronbach Alpha value in this study was found to be 0.896.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Bakircay University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No